CLINICAL TRIAL: NCT06467617
Title: A Phase II Clinical Study of Adabrelimab Combined With Carboplatin, Albumin-bound Paclitaxel, and Recaticimab in Perioperative Treatment of Resectable NSCLC
Brief Title: Adebrelimab Plus Chemo and Recaticimab in Perioperative Treatment of Resectable NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Chest Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Jinghui Wang, Director of Research Laboratory, Beijing Chest Hospital, Beijing Chest Hospital, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJXK-2024-IIT-05
Record Dates: First submitted 2024-06-13; First posted 2024-06-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab plus albumin-bound paclitaxel, carboplatin and recaticimab (Experimental): Participants will receive Adebrelimab 1200mg IV on Day 1 of a 21-Day cycle plus albumin-bound paclitaxel 260 mg/m2, IV, divided by D1,8 of a 21-Day cycle plus Carboplatin AUC 5mg/mL/min, IV, and recaticimab 150 mg, SC on the Day 1 of a 21-Day cycle
  Interventions: Drug: Adebrelimab plus albumin-bound paclitaxel, carboplatin and recaticimab

INTERVENTIONS:
Drug: Adebrelimab plus albumin-bound paclitaxel, carboplatin and recaticimab — Adebrelimab (1200 mg,IV, D1, Q3W) +
  albumin-bound paclitaxel (260 mg/m2, IV, divided by D1,8,Q3W) +
  carboplatin (AUC 5mg/mL/min, IV, D1,Q3W) +
  recaticimab (150 mg, SC, D1,Q3W)
  21-day cycle

SUMMARY:
Current studies confirmed that the immune perioperative treatment with combination chemotherapy curative effect and safety of resectable NSCLC, but its short-term curative effect and long-term survival benefit remains to be further improved to explore the new way of immune combination therapy.

Experimental study showed that the inhibition of PCSK9 could significantly increase in tumor cells of the immune response in mice, inhibit the PCSK9 enhanced anti-tumor immune response of mice can be further coordinate with immune checkpoint therapy, forming a lasting anti-tumor immune effect.

There are no reports on the peri-operative treatment of immune combined with chemotherapy and PCSK-9 inhibitors in patients with resectable NSCLC.

Based on the above, the aim of this study is to explore the efficacy and safety of Adebrelimab combined with recaticimab and chemotherapy in the perioperative treatment of patients with resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male and female;
2. ECOG PS 0-1;
3. Histologically or cytologically confirmed operable stage II-III NSCLC (stages II, IIIA, and T3N2M0 IIIB) according to the UICC and AJCC 8th edition TNM staging system. Non-massive metastases (short diameter ≤2cm Lymph nodes) with expected complete resectable N2;
4. With a measurable lesions (per RECIST 1.1 standard, tumor lesions on CT scan length to diameter 10 mm, or lymph node lesions on CT scans short diameter 15 mm or higher);
5. Anti-tumor treatment (radiotherapy, chemotherapy, surgery, and targeted therapy) naive enrollment;
6. Enough of lung function to go through R0 resection with a purpose of cure;
7. Normal main organs function, should meet the following criteria: (1) the blood routine examination shall meet within 14 days (without blood transfusion, hematopoietic factor not used and unused drugs to correct) a. ANC≥1.8 x 109 / L; B. Hb≥100 g/L; C. PLT ≥ 125×109/L; (2) Biochemical examination must meet the following criteria: a. TBIL ≤ 1.5ULN; B. ALT、AST≤2.5 ULN; Serum creatinine sCr≤1.5ULN, endogenous creatinine clearance≥50ml/min (Cockcroft-Gault formula)

Exclusion criteria

1. Known EGFR or ALK mutation;
2. T4 tumors invading the heart, great vessels, trachea, recurrent laryngeal nerve, esophagus, vertebral body, tracheal carina, Upper sulcus lung cancer;
3. Use of immunosuppressive drugs within 4 weeks before the first dose of study drug, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (i.e., ≤10 mg/day of prednisolone or other corticosteroids at physiological doses of equivalent drugs, with discontinuation of the drug for ≥1 week);
4. Received immunoregulatory effects of herbal medicine or Immune regulating effect of drugs (including thymosin, interferon, interleukin, except for local control Pleural effusion use) within 4 weeks before the first use of the study drug;
5. Malignant tumors other than NSCLC occurred within 5 years before enrollment.
6. Administered Live attenuated vaccine ≤ 4 weeks before the first dose or will be planned for the duration of the study；
7. Current are participating in clinical research and treatment of intrusive, or within 4 weeks before the first delivery received study drugs or other treatments; Not fully recovered from any intervention-related toxicity and/or complications before the first dose (i.e., ≤ grade 1 or baseline, excluding fatigue or alopecia)；
8. Severe infection (e.g., requiring intravenous antibiotics, antifungal or antiviral drugs) within 4 weeks before the first dose, or unexplained fever during screening/before the first dose. 38.5°C；
9. Have or suspected a history of pneumonia/interstitial lung disease or any lung disease that would interfere with pulmonary function testing;
10. With any active history of autoimmune disease or autoimmune diseases; Patients with complete remission of childhood asthma without any intervention in adulthood or with vitiligo were eligible;
11. With congenital or acquired immune function defects, such as human immunodeficiency virus (HIV) infection, active hepatitis B, hepatitis C, hepatitis B and hepatitis C infection together and alcoholic liver cirrhosis patients;
12. Patients with grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥450ms in men and ≥470ms in women). According to NYHA standard, grade III ~ Ⅳ cardiac insufficiency, or heart colour to exceed examination prompt left ventricular ejection fraction (LVEF) < 50% into the group of the first six months happened myocardial infarction, heart failure, New York heart association class II or above has not been control angina pectoris, out of control of severe ventricular arrhythmia, with clinical significance of cardiac disease, Or abnormal electrocardiogram (ecg) indicate that acute ischemia or active conduction system;
13. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) more than 2 times the upper limit of normal value, or total bilirubin more than 1.5 times the upper limit of normal value (ULN); Creatine kinase (CK) was more than 3 times the upper limit of normal; There were major hemorrhagic events or arteriovenous thrombotic events
14. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
15. Known allergy, hypersensitivity, or intolerance to the study drug or its excipients;
16. Any condition considered by the investigator to be present that could harm the subject or cause the subject to be unable to meet or perform the requirements of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
pCR | 1.5 year
  Pathological complete response；

SECONDARY OUTCOMES:
MPR | through study completion, an average of 2 year
  major pathologic response
ORR | through study completion, an average of 2 year
  Objective response rate
EFS | through study completion, an average of 2 year
  Event free survival
DFS | through study completion, an average of 2 year
  Disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jinghui Wang, Study Chair — Director of Research Laboratory, Beijing Chest Hospital
Locations (1):
- Beijing Chest Hospital, Beijing, Beijing Municipality, China